CLINICAL TRIAL: NCT07200076
Title: Comparison of Mean Duration of Post Operative Analgesia Following QL-2 Block vs QL-3 Block Using Ropivacain 0.25% in Patients Undergoing Unilateral Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Dr Muhammad Ayaz, Principal investigator, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BVH-2025-CT-010
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Inguinal Hernia Unilateral
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QLB-2 (posterior QL block) Group (Active Comparator)
  Interventions: Procedure: Quadratus Lumborum (QL) Block
- QLB-3 (transmuscular QL block) Group (Active Comparator)
  Interventions: Procedure: Quadratus Lumborum (QL) Block

INTERVENTIONS:
Procedure: Quadratus Lumborum (QL) Block — In the QLB-2 approach, a needle will be inserted in-plane from anterior to posterior, directed towards the posterior QL muscle border, and a 20 ml solution of 0.25% ropivacaine will be injected.
  For the QLB-3 approach, the needle will be inserted in-plane from anterior to posterior, traversing the QL muscle's proper fascia to target the plane between the QL and PM muscles, and a 20 ml solution of 0.25% ropivacaine will be injected.

SUMMARY:
To compare the mean dulation of post operative analgesia following QL2 block (posterior quadratus lumborum block) and the QL3 block (transmuscular quadratus lumborum block) using ropivacaine 0.25% in patients undergoing unilateral inguinai hernia repair.

Rationale of the proposed study is to find an optimal approach for quadratus lumborum block (QLB) in the context of local population as no local study has already been carried out for our population. The study seeks to determine which approach provides superior postoperative pain relief and aspires to establish a clear rationale for the application of one technique over the other in local population. By uncovering the strengths and limitations of each approach, the study intends to guide local clinicians in making informed decisions for optimizing postoperative pain management strategies. The outcomes of this study are anticipated to have a substantial impact on clinical practice, potentially leading to improved patient outcomes, reduced opioid consumption, and enhanced patient comfort following inguinal hernia repair surgeries in local settings.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years ASA status 1 or 2 Scheduled for unilateral inguinal hernia repair under General Anaesthesia

Exclusion Criteria:

* Patient refusal Patients with pre-existing coagulation abnormalities INR more thnn 1.5 Patients with Strangulated hernia Hypersensitivity to local anaestiretics. Local infection at procedure sito.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change in systolic Blood pressure | Baseline, 30 minutes, 2 hours, 4 hours, 8 hours, 12 hours 24 hours
Mean duration of analgesia | Baseline, 30 minutes, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours
  assessed using the Visual Analog Score (VAS) ranging tiom 0-10 (0= no pain, l0= the most severe unbearable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No